CLINICAL TRIAL: NCT00505024
Title: A Randomized Clinical Trial of the Efficacy of an Interactive Voice Response System (IVRS) for Managing Symptoms of Patients Following Thoracic Surgery
Brief Title: Interactive Voice Response System (IVRS) for Managing Symptoms of Patients Following Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-0299
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Cancer; Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Esophageal Cancer; Lung Cancer; Interactive Voice Response System; IVRS
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVRS Only (Experimental)
  Interventions: Behavioral: Interactive Voice Response System
- IVRS + Symptoms Report (Experimental)
  Interventions: Behavioral: Interactive Voice Response System; Other: Symptoms Report

INTERVENTIONS:
Behavioral: Interactive Voice Response System — Calls twice weekly, where the system will ask you to rate types of symptoms on a scale from 0 to 10.
  Other Names: IVRS
Other: Symptoms Report — A report of severe symptoms will be sent to your doctor or nurse.
  Arms: IVRS + Symptoms Report

SUMMARY:
To test the effectiveness of the interactive voice response telephone system with a triage/feedback component that incorporates timely symptom assessment, feedback to physicians, critical treatment guidelines for managing selected symptoms (distress, sleep disturbance, shortness of breath, constipation, and pain) in a cohort of cancer patients during the first month post-thoracic surgery.

This interactive voice response system (IVR) will be evaluated in a randomized clinical trial with an intervention group (IVR symptom assessment with triage) and a control group (IVR symptom assessment only).

We hypotheses that:

1. Patients in the MDASI-IVR plus triage group will have less symptom burden (less symptom severity, less symptom related interference, and better satisfaction of symptom control, better physical and emotional well-being) over the month of the trial compared to the control group.
2. Patients in the MDASI-IVR plus triage group will have more frequent documentation of symptom management in line with treatment guidelines compared to the control group.

DETAILED DESCRIPTION:
The IVRS is a special telephone system that calls patients and asks questions about symptoms. The system can record and report severe symptoms to a patient's doctor by e-mail, fax, or pager. All patients are encouraged to report and discuss any severe symptoms to your treating clinicians.

If you agree to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. Participants in one group will complete symptom surveys on the IVRS. Participants in the other group will complete symptom surveys on the IVRS, and (in addition) a report of severe symptoms will be sent to their doctor or nurse.

All participants will initially be asked to complete 2 surveys (before surgery) that will ask about any symptoms you may be having and your general quality of life. It will take about 10 minutes to complete both surveys. You will also be asked to provide some demographic information, such as your age, gender, employment status, and ethnicity.

Before you are discharged from the hospital (after your surgery), a member of the study staff will visit you and teach you how to use the IVRS system, and you will then continue participation according to your assigned group.

After you are discharged from the hospital, the system will be set up to call you (all participants) twice a week until 1 month after your surgery. It will be automated to ask you to rate 14 types of symptoms (such as pain, fatigue, nausea, sleep disturbance and 6 other items, such as how your symptoms interfere with your day-to-day activity, mood, and enjoyment of life) on a scale from 0 to 10. Zero (0) means that the symptom is not present, and 10 means that you are experiencing the symptom at its worst. The call should last from 3-5 minutes. For participants in the other group, a symptom report will also be sent to your doctor or nurse.

One month after surgery, you will have a phone call from a member of the research staff. During this phone call, you will be asked to provide additional information about the symptoms you experienced and how you managed them.This phone call will last about 20 minutes. If you are not able to be reached by research staff the first time you are called, you will be called again at another time between the 5th and 6th week after your surgery.

THIS IS AN INVESTIGATIONAL STUDY. Up to 130 patients (65 in each group) will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for thoracic surgery for NSCLC, esophageal cancer and lung metastasis
2. Patients 18 years of age or older
3. Men and women of all ethnic groups who are English-speaking, and
4. Patients residing in the United States. (The IVR system is not yet available in other languages. The United States residency requirement (MDACC is an international referral center) will allow us to follow patients for the duration of the study.)

Exclusion Criteria:

1. Patients with a current diagnosis of psychosis or dementia
2. Patients who have difficulty understanding the intent of the study
3. Patients who cannot complete the assessment tools independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To study the effectiveness of the interactive voice response system (IVRS), which is designed to send a report to a patient's doctor about severe symptoms they are experiencing. | 3 Years

SECONDARY OUTCOMES:
To study if systematic symptom assessment (by the use of IVRS) is another way to report symptoms rather than the usual method, which is calling the doctor when there is a problem. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org